CLINICAL TRIAL: NCT06146556
Title: Concealed Myocardial Abnormalities by Cardiac Magnetic Resonance Imaging in Idiopathic Ventricular Arrhythmias
Brief Title: Concealed Myocardial Abnormalities by Cardiac Magnetic Resonance Imaging in Idiopathic VT
Status: Active, not recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Abdallah Hasaballah Farag, Assistant lecturer, Assiut University
Other Study IDs: Idiopathic VT imaging
Record Dates: First submitted 2023-09-22; First posted 2023-11-24 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Premature Ventricular Contractions
Keywords: idiopathic VAs
MeSH Terms: conditions — Ventricular Premature Complexes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: catheter based ablation — electrophysiological catheter based ablation of ventricular arrhythmia

SUMMARY:
Idiopathic Ventricular arrhythmia (VAs) refers to VAs that occur in the absence of clinically apparent structural heart disease. The outflow tracts (OTs) are the most common origin of idiopathic VAs and PVCs, accounting for approximately 10% of all patients referred for evaluation of VAs with the RVOT being the origin of about 70-80% of these arrhythmias.

Studies have shown that increased PVC burden was associated with reduced LV function, a higher incidence of heart failure, and a higher risk of death.

The diagnosis, prognostication and treatment of patients with VAs are challenging. A routine diagnostic workup that includes transthoracic echocardiography and an assessment for the presence of coronary artery disease (CAD) as recommended by current clinical guidelines cannot recognize focal structural abnormalities or underlying structural heart disease (SHD) in a substantial proportion of patients. Cardiac magnetic resonance (CMR) provides an excellent assessment of cardiac morphology and function and enables a detailed myocardial tissue characterization with a high degree of precision. CMR is widely regarded as the gold standard for identifying structural arrhythmogenic substrates in patients with VAs and normal echocardiography.

DETAILED DESCRIPTION:
Idiopathic Ventricular arrhythmia (VAs) refers to VAs that occur in the absence of clinically apparent structural heart disease. The outflow tracts (OTs) are the most common origin of idiopathic VT and PVCs, accounting for approximately 10% of all patients referred for evaluation of VT with the RVOT being the origin of about 70-80% of these arrhythmias.

Studies have shown that increased PVC burden was associated with reduced LV function, a higher incidence of heart failure, and a higher risk of death.

The diagnosis, prognostication and treatment of patients with VAs are challenging. A routine diagnostic workup that includes transthoracic echocardiography and an assessment for the presence of coronary artery disease (CAD) as recommended by current clinical guidelines cannot recognize focal structural abnormalities or underlying structural heart disease (SHD) in a substantial proportion of patients. Cardiac magnetic resonance (CMR) provides an excellent assessment of cardiac morphology and function and enables a detailed myocardial tissue characterization with a high degree of precision. CMR is widely regarded as the gold standard for identifying structural arrhythmogenic substrates in patients with VAs and normal echocardiography. More importantly, myocardial structural abnormalities detected on CMR in patients with idiopathic VAs are associated with an increased risk of arrhythmic events and worse clinical outcomes.

However, little is known regarding the added value of CMR including feature-tracking strain CMR (FT-CMR) in identifying underlying myocardial abnormalities and biventricular dysfunction in a relatively 'healthy' population of patients with VAs and normal echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* All patients presented with idiopathic ventricular arrhythmias with normal diagnostic routine workup at Assiut university heart hospital. Diagnostic work up including a normal ECG with no changes suggestive of structural heart disease, normal echocardiography ﬁndings and no evidence of CAD on either invasive or non-invasive imaging

Exclusion Criteria:

* (1) known history of cardiac disease (CAD, cardiomyopathy, congenital heart disease, more than mild valvular disease, previous cardiac surgery of any type), any severe systemic disease with cardiac involvement.

  (2) Allergy to gadolinium-based contrast agents, an estimated glomerular ﬁltration rate < 30 mL/min/1.73 m2.

  (3) Any contraindication to the MR environment (e.g., MR-unsafe implants/devices, shrapnel injury), pregnancy and claustrophobia

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients presented with idiopathic ventricular arrhythmias with normal diagnostic routine workup at Assiut university heart hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess the diagnostic yield of cardiac MRI in early detection of biventricular dysfunction in patients with idiopathic VAs | one year
  the value of CMR in evaluation of ventricular dysfunction in patients with ventricular arrhythmias

SECONDARY OUTCOMES:
Assess the clinical predictors of myocardial dysfunction | one year
  different risk factors for ventricular dysfunction including demographic data, clinical data as regards age, diabetus mellitus, hypertension, family history
Assess the PVCs burden association with myocardial abnormalities | one year
  Premature ventricular ectopics burden associated with myocardial abnormalities as detected by ECG Holter monitoring as regard frequency of ectopics
Assess the PVCs morphology association with myocardial abnormalities | one year
  assess PVCs morphology in holter monitoring as left or right bundle branch block morphology and axis

CONTACTS AND LOCATIONS:
Overall Officials: shimaa sayed, MD, Principal Investigator — Lecturer of cardiovascular medicine
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] 1.Aliot EM, Stevenson WG, Almendral-Garrote JM, Bogun F, Calkins CH, Delacretaz E, et al. EHRA/HRS expert consensus on catheter ablation of ventricular arrhythmias. Vol. 11, Europace. 2009. p. 771-817 2.Kim YH, Chen SA, Ernst S, Guzman CE, Han S, Kalarus Z, et al. 2019 APHRS expert consensus statement on three-dimensional mapping systems for tachycardia developed in collaboration with HRS, EHRA, and LAHRS. Vol. 36, Journal of Arrhythmia. Wiley-Blackwell; 2020. p. 215-70. 3..Pedersen CT, Kay GN, Kalman J, Borggrefe M, Della-Bella P, Dickfeld T, et al. EHRA/HRS/APHRS expert consensus on ventricular arrhythmias. EP Europace 2014 Sep 1. Available from: https://dx.doi.org/10.1093/europace/euu194 4.Andreini D, Dello Russo A, Pontone G, Mushtaq S, Conte E, Perchinunno M, et al. CMR for Identifying the Substrate of Ventricular Arrhythmia in Patients With Normal Echocardiography. Cardiovascular Imaging . 2020 Feb 1 https://www.jacc.org/doi/10.1016/j.jcmg.2019.04.023 5.Muser D, Santangeli P, Castro SA, Casado Arroyo R, Maeda S, Benhayon DA, et al. Risk Stratification of Patients With Apparently Idiopathic Premature Ventricular Contractions: A Multicenter International CMR Registry. JACC Clin Electrophysiol. 2020 Jun 1;6(6):722-35